CLINICAL TRIAL: NCT00247455
Title: Long-term Effect of Cereal Fibre on Abdominal Fat in Insulin Resistant Subjects
Brief Title: Fibre and Appetite Regulation Trial (FART)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Diabetes Association (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDA1323; Can Diabetes Assoc Grant 1323; CIHR Grant OOP-64648
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2007-08

CONDITIONS: Obesity; Diabetes
Keywords: Human nutrition; Dietary fibre; Insulin resistance; Obesity; Glucose; Colonic fermentation; Short chain fatty acids; GLP-1; Appetite; Abdominal fat
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Low fibre breakfast cereal (puffed rice/cornflakes)
Drug: High fibre cereal (All Bran/Bran Flakes)

SUMMARY:
High intake of cereal fibre has been shown to be associated with reduced weight gain and improved insulin sensitivity. We hypothesize these effects are due to the short chain fatty acids derived from the bacterial fermentation (breakdown) of fibre in the colon (large intestine). Insulin resistant subjects will be randomized to receive 2 servings of a low-fibre cereal (eg. puffed rice) or 2 servings of a high-fibre cereal (wheat bran cereal) per day for one year. The effects of the diets on body weight, appetite, abdominal fat, blood short chain fatty acids, glucose, insulin, lipids and hormones will be measured

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic male or non-pregnant females
* aged 18-60
* BMI<36
* fasting insulin >40pmol/L (70%ile)

Exclusion Criteria:

* intention to lose >5kg in weight
* presence of diabetes (fasting glucose >6.9mmol/L)
* use of diuretics, beta-blockers or weight reducing drugs
* use of antibiotics in last 3 months and use of antibiotics more than once annually for the last 2 years
* significant gastrointestinal, liver or kidney disease
* use of lipid-lowering drug
* major medical or surgical event in last 6 mo.
* fibre intake >30g/d
* inability to eat low or high fibre breakfast cereals
* unwilling or unable to give consent or comply with protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2002-03; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Serum acetate concentration | 0, 3, 6, 9 and 12 months
Serum butyrate concentration | 0, 3, 6, 9 and 12 months
Plasma GLP-1 concentration | 0, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Fasting glucose and insulin | 0, 3, 6, 9 and 12 months
HOMA insulin resistance and beta cell function | 0, 3, 6, 9 and 12 months
postprandial glucose and insulin | 0, 3, 6, 9 and 12 months
Body weight | 0, 3, 6, 9 and 12 months
waist circumference | 0, 3, 6, 9 and 12 months
Abdominal fat | 0 and 12 months
food intake | 0, 3, 6, 9 and 12 months
Fasting lipids (cholesterol, triglyceride, HDL, LDL) | 0, 3, 6, 9 and 12 months
Fasting and postprandial free fatty acids and triglycerides | 0, 3, 6, 9 and 12 months
Fasting and postprandial c-peptide | 0, 3, 6, 9 and 12 months
C-peptide/insulin ratio as marker of hepatic insulin extraction | 0, 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, BM, BCh, PhD, DM, Principal Investigator — University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Freeland KR, Wilson C, Wolever TM. Adaptation of colonic fermentation and glucagon-like peptide-1 secretion with increased wheat fibre intake for 1 year in hyperinsulinaemic human subjects. Br J Nutr. 2010 Jan;103(1):82-90. doi: 10.1017/S0007114509991462. Epub 2009 Aug 7. PMID 19664300